CLINICAL TRIAL: NCT06019065
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AJA001 in Fasting and Fed Healthy Participants
Brief Title: A SAD, MAD and Food Effect Study to Evaluate the Safety, Tolerability, PK, and PD of AJA001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AJNA Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AJA001-001
Record Dates: First submitted 2023-08-11; First posted 2023-08-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (16):
- Cohort A1: Single ascending dose of AJA001 (Experimental): AJA001 active q.d. 2.2 mL oral dose level 1
  Interventions: Drug: AJA001
- Cohort A1: Single ascending dose of placebo (Placebo Comparator): AJA001 placebo q.d. 2.2 mL oral dose level 1
  Interventions: Other: Placebo
- Cohort A2: Single ascending dose of AJA001 (Experimental): AJA001 active q.d. ascending oral dose level 2
  Interventions: Drug: AJA001
- Cohort A2: Single ascending dose of placebo (Placebo Comparator): AJA001 placebo q.d. ascending oral dose level 2
  Interventions: Other: Placebo
- Cohort A3: Single ascending dose of AJA001 (Experimental): AJA001 active q.d. ascending oral dose level 3
  Interventions: Drug: AJA001
- Cohort A3: Single ascending dose of placebo (Placebo Comparator): AJA001 placebo q.d. ascending oral dose level 3
  Interventions: Other: Placebo
- Cohort A4: Single ascending dose of AJA001 (Experimental): AJA001 active q.d. ascending oral dose level 4
  Interventions: Drug: AJA001
- Cohort A4: Single ascending dose of placebo (Placebo Comparator): AJA001 placebo q.d. ascending oral dose level 4
  Interventions: Other: Placebo
- Cohort B1: Multiple ascending doses of AJA001 (Experimental): AJA001 active b.i.d. oral dose level 1
  Interventions: Drug: AJA001
- Cohort B1: Multiple ascending doses of placebo (Placebo Comparator): AJA001 placebo b.i.d. oral dose level 1
  Interventions: Other: Placebo
- Cohort B2: Multiple ascending doses of AJA001 (Experimental): AJA001 active b.i.d. oral dose level 2
  Interventions: Drug: AJA001
- Cohort B2: Multiple ascending doses of placebo (Placebo Comparator): AJA001 placebo b.i.d. oral dose level 2
  Interventions: Other: Placebo
- Cohort B3: Multiple ascending doses of AJA001 (Experimental): AJA001 active b.i.d. oral dose level 3
  Interventions: Drug: AJA001
- Cohort B3: Multiple ascending doses of placebo (Placebo Comparator): AJA001 placebo b.i.d. oral dose level 3
  Interventions: Other: Placebo
- Cohort B4: Multiple ascending doses of AJA001 (Experimental): AJA001 active b.i.d. oral dose level 4
  Interventions: Drug: AJA001
- Cohort B4: Multiple ascending doses of placebo (Placebo Comparator): AJA001 placebo b.i.d. oral dose level 4
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AJA001 — AJA001
  Arms: Cohort A1: Single ascending dose of AJA001; Cohort A2: Single ascending dose of AJA001; Cohort A3: Single ascending dose of AJA001; Cohort A4: Single ascending dose of AJA001; Cohort B1: Multiple ascending doses of AJA001; Cohort B2: Multiple ascending doses of AJA001; Cohort B3: Multiple ascending doses of AJA001; Cohort B4: Multiple ascending doses of AJA001
Other: Placebo — Placebo
  Arms: Cohort A1: Single ascending dose of placebo; Cohort A2: Single ascending dose of placebo; Cohort A3: Single ascending dose of placebo; Cohort A4: Single ascending dose of placebo; Cohort B1: Multiple ascending doses of placebo; Cohort B2: Multiple ascending doses of placebo; Cohort B3: Multiple ascending doses of placebo; Cohort B4: Multiple ascending doses of placebo

SUMMARY:
This is a Phase 1, double-blind, randomized, placebo- controlled, SAD and MAD study to assess safety, tolerability, PK, and PD of AJA001 in fasted healthy participants. Food effect will be evaluated in one cross-over SAD fed dose cohort.

DETAILED DESCRIPTION:
The study is comprised of two parts, Part A (SAD) and Part B (MAD). Participants will be randomized (active or placebo) in each cohort of Parts A and B. Participants in Part A will receive a single dose of AJA001 or placebo on Day 1. Part A will include a fed-cohort (A-X) for one cohort where the participants will return to the clinical site on Day 14 to receive AJA001 or placebo. Participants in Part B will receive a split dose of AJA001 or placebo, where one dose will be administered as two equal doses taken twice daily, (BID; administered approximately every 12 hours [± 30 minutes]) for 6 consecutive days (Day 1-Day 6), and 1 morning dose on Day 7.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed ethics committee (EC)-approved consent form prior to any study procedures, can understand and comply with the requirements of the study, and are able to communicate with the Investigator
2. Males and females, aged 18 and 65 years (inclusive), with body mass index (BMI) of 18 32.0 kg/m2 and body weight ≥50.0 kg at screening
3. No known allergic reaction to cannabis products and formulation components (Glyceryl Monolinoleate, NF and organic chocolate mint flavoring agent)
4. Medically healthy with no clinically significant medical history (fully resolved childhood asthma and mild asthma that does not require a reliever more than once per month, and does not require a preventer or any additional therapies is not considered clinically significant and permissible), physical examination, laboratory profiles, vital signs, or ECG, as deemed by the Investigator
5. Must have hepatic and renal clinical laboratory test results (ALT, AST, total bilirubin [including direct and indirect bilirubin results], and eGFR) within a laboratory defined normal range
6. Male participants who are not vasectomized for at least 6 months prior to dosing and who are sexually active with a female partner of childbearing potential must be willing to use one of the acceptable contraceptive methods specified below under "Contraception" in Section 8.1 from the first dose and for 90 days after the last dose
7. Females of childbearing potential who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomized at least 6 months prior to the first study drug administration) must be willing to use one of the acceptable contraceptive methods specified below specified below under "Contraception" throughout the study and for at least 3 months after the last study drug administration
8. Refrain from donating sperm for the duration of the study and for at least 90 days after the last dose of investigational product (IP)
9. Females must have a negative serum pregnancy test (SPT) at screening and urinary pregnancy test (UPT) at check-in on Day -1
10. Agree to frequent blood sampling during the course of the study and with adequate venous access
11. Agree to be confined for parts of the study in the Phase 1 unit and follow study procedures
12. Agree to comply with the study-specified diet while confined in the Phase 1 unit. Participants in the Part A - cohort which enter the fed cross-over design (A-X) must agree to complete consumption of a standardized high-fat breakfast during the fed period on Day 15
13. Negative drug and alcohol tests at screening and at admissions on Day -1 and willing to abstain from alcohol/illegal drug use from the screening visit until the End of Study (EOS) visit
14. Able to read, understand, provide signed informed consent, communicate adequately, and comply with the requirements for the entire study.

Exclusion Criteria:

1. Use of any medications or over the-counter (OTC) products within 10 days or 5 half lives (whichever is longer) prior to administration of study medication (including analgesics [note: except paracetamol up to 2 g per day], antibiotics, hormonal contraceptives* [except, which is permitted], natural food supplements, vitamins, garlic as a supplement)

   *Note: Stable doses of oral contraceptives for birth control in women of childbearing potential (WOCBP) (minimum of 3 months without issue as deemed by the Investigator) will be allowed. No other hormonal treatment will be allowed.
2. Use of an investigational drug or participation in an investigational study within 30 days (or 5 half-lives of the investigational drug, whichever is longer) prior to dosing
3. Use of known inhibitors or inducers of hepatic drug metabolism (e.g., rifampin, carbamazepine, phenytoin, norethindrone, barbiturates [e.g., phenobarbital], dexamethasone, antidepressants [e.g., fluoxetine, paroxetine], proton pump inhibitors, ketoconazole) 1 month before the start of the study (Day 1)
4. Hypersensitivity or any significant allergic reaction to the investigational compound/compound class being used in this study or any ingredients of this medication
5. Medical history or any clinically significant disorder (as determined by the Investigator and Sponsor) including but not limited to: clinically significant allergies, asthma (fully resolved childhood asthma with no reoccurrences in adulthood is permissible), angioedema, pulmonary, bronchospasm, ulcer disease, gastrointestinal (GI), GI bleeding, coagulation defects, hypertension, edema, heart failure, hypokalemia, cardiovascular disease, significant dermatologic diseases or conditions; hematological, neurological, psychiatric, hepatic, or renal disorders; condition that would significantly influence the immune response; or history of infections of unexplained frequency or severity;
6. Personal diagnosis or first-degree relative diagnosis of psychosis/schizophrenia
7. Presence of current psychiatric condition, suicide ideations or psychiatric condition requiring pharmacological management within the last 6 months
8. History or presence of any condition that, in the opinion of the Investigator, could interfere with the study conduct or observation (to be confirmed by medical history)
9. Has used any tobacco / nicotine-containing products (e.g., cigarettes, vaporizers, cigars, pipe tobacco, smokeless tobacco, nicotine gum, lozenges, patches) on more than 5 occasions within 1 month of the Screening visit
10. History of significant drug abuse within 1 year prior to screening or use of drugs such as cannabis within 2 months prior to the screening visit or drugs such as cocaine, phencyclidine (PCP), crack, opioid derivatives including heroin, and amphetamine derivatives within 1 year prior to screening.
11. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit that exceeds 14 units of alcohol per week for female participants and 21 units for male participants (1 unit = 150 mL of wine, 375 mL of mid strength beer, or 30 mL of distilled alcohol 40%).
12. History of or risk for seizures (one-off febrile seizure as a child is permissible)
13. History or positive screening results to hepatitis B surface antigen or C virus Ab tests, or to human immunodeficiency virus (HIV) Ag/Ab combination, or has known immune deficiency disease at screening
14. Surgical (history of stomach or intestinal surgery or resection) or medical condition (evidence of prior chronic GI disease such a cholecystitis, cholecystectomy, Gilbert's syndrome) that would interfere with gastric motility, pH, or absorption of study drug
15. Laboratory values outside normal ranges based on the laboratory reference values and are clinically significant or ≥ Grade 1 Common Terminology Criteria for Adverse Events (CTCAE; v5.0) (repeat testing is allowed once) at screening and Day -1
16. Presence of out-of-range cardiac interval (PR ≥120 msec, PR ≤220 msec, QRSD <120 msec and QTcF ≤450 msec for males and females) on the ECG at screening and Day -1 or other clinically significant ECG abnormalities, unless deemed non significant by the Investigator
17. Presence of clinically significant vital sign abnormalities (systolic BP lower than 90 or over 140 mmHg, diastolic BP lower than 40 or over 90 mmHg, HR less than 40 or over 100 bpm, or RR less than 10 or over 22 resp/min) at screening and Day -1.
18. Use of Δ9-tetrahydrocannabinol (THC)- or cannabidiol (CBD)-containing products within 60 days of start of study (Day 1)
19. Serious illness in the 30 days preceding the beginning of treatment on Day 1 (i.e., that resulted in hospitalization)
20. Receipt of treatment for any type of internal cancer within the 5 years prior to enrollment (fully treated and resolved basal cell carcinoma and or squamous cell carcinoma are permissible)
21. Females who are pregnant, plan to become pregnant during the study, or are breastfeeding a child
22. Positive alcohol breath test or urine drug screen at screening or at admissions on Day -1
23. Blood or plasma donation (500 mL) within the past month, or receipt of blood transfusion within 1 month prior to Day 1
24. Employee, family member, or student of the Investigator or clinical site(s)

Contraception:

Male participants who are not vasectomized for at least 6 months prior to dosing, and who are sexually active with a female partner of childbearing potential must be willing to use one of the following acceptable contraceptive methods from the first dose and for 90 days after the last dose:

* Simultaneous use of condom and established use of oral, injected or implanted hormonal contraceptive (at least 4 weeks prior to screening)
* Simultaneous use of condom and placement of intrauterine device (IUD) or intrauterine system (IUS)

There are no contraceptive requirements if any of following conditions apply:

* Sexual partner is surgically sterile;
* Partner of non-childbearing potential;
* Same sex relationship;
* Abstinence from heterosexual intercourse as usual and preferred lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.

Females of childbearing potential who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomised at least 6 months prior to the first study drug administration) must be willing to use one of the following acceptable contraceptive methods throughout the study and for at least 3 months after the last study drug administration:

- Simultaneous use of intrauterine contraceptive device without hormone release system placed at least 4 weeks prior to the first study drug administration; or intrauterine contraceptive device with hormone release system placed at least 12 weeks prior to first study drug administration; or oral hormonal contraceptives (minimum 12 week use without issue), and a condom for the male partner.

Females of non-childbearing potential must be:

* Post-menopausal (absence of menses for at least 12 months prior to the first study drug administration) with confirmation of the post menopausal status by documented FSH level ≥40 mIU/mL; or
* Surgically sterile (complete hysterectomy or bilateral oophorectomy at least 3 months prior to the first study drug administration).

Please note women with tubal ligation will be required to undergo a pregnancy tests and partner to use a condom (ie. they will be treated as WOCBP).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 21 days
  Incidence, severity and relationship of Adverse events (AEs)
Serious Adverse Events | Up to 21 days
  Incidence of Serious adverse events (SAEs)
Adverse Events of Special Interest | Up to 21 days
  Incidence of AEs of special interest (AESI), including abnormal clinically significant liver function test values (aspartate aminotransferase, alanine aminotransferase, total bilirubin and estimated glomerular filtration rate) due to major active pharmaceutical ingredient
Changes from baseline in hematology | Up to 21 days
  Number of participants with changes from baseline in hematocrit, hemoglobin, mean cell hemoglobin, mean cell hemoglobin concentration, mean cell volume, platelet count, red blood cell count, reticulocyte count, white blood cell count, and differential white blood cell count
Changes from baseline in serum chemistry | Up to 21 days
  Number of participants with changes from baseline in aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma glutamyl transferase, sodium, potassium, chloride, calcium, magnesium, phosphorus, glucose, serum urea, uric acid, total bilirubin, creatinine, total protein, albumin, total cholesterol, triglycerides, creatinine phosphokinase, and follicle-stimulating hormone
Changes from baseline in urinalysis | Up to 21 days
  Number of participants with changes from baseline in microscopic examination, specific gravity, pH, protein, glucose, ketones, blood, urobilinogen, bilirubin, nitrites, leucocytes, immunoassay for THC
Changes from baseline in blood pressure | Up to 21 days
  Number of participants with changes from baseline in systolic and diastolic blood pressure in mm Hg
Changes from baseline in heart rate | Up to 21 days
  Number of participants with changes from baseline in pulse rate (beats/minute)
Changes from baseline in respiratory rate | Up to 21 days
  Number of participants with changes from baseline in respiratory rate (breaths/minute)
Changes from baseline in body temperature | Up to 21 days
  Number of participants with changes from baseline in body temperature (tympanic; °C)
Changes from baseline in ECG recording of heart rate | Up to 21 days
  Number of participants with changes in 12-lead electrocardiogram (ECG) recordings of heart rate in beats/minute
Changes from baseline in ECG recording of PR interval | Up to 21 days
  Number of participants with changes in 12-lead electrocardiogram (ECG) recordings of PR interval in msec
Changes from baseline in ECG recording of RR interval | Up to 21 days
  Number of participants with changes in 12-lead electrocardiogram (ECG) recordings of RR interval in msec
Changes from baseline in ECG recording of QRS duration | Up to 21 days
  Number of participants with changes in 12-lead electrocardiogram (ECG) recordings of QRS duration in msec
Changes from baseline in ECG recording of QT interval | Up to 21 days
  12-lead electrocardiogram (ECG) recordings of QT interval in msec
Changes from baseline in ECG recording of QTcF | Up to 21 days
  Number of participants with changes in 12-lead electrocardiogram (ECG) recordings of QTcF in msec
Clinically significant physical examination findings | Up to 21 days
  Number of participants with changes in the following parameters assessed during physical exams: general appearance, head, ears, eyes, nose, throat, neck (including thyroid), skin, cardiovascular system, respiratory system, gastrointestinal system, musculoskeletal system, lymph nodes and nervous system
Changes in suicidal ideation and behavior | Up to 21 days
  Number of participants with changes in Columbia Suicide Severity Rating Scale evaluation of suicidal ideation (yes/no), intensity of ideation (1-5 with 1 being the least severe and 5 being the most severe), and suicidal behavior (yes/no; if yes, include the number of attempts)
Use of concomitant medications | Up to 21 days
  All medications taken after the first dose of the study drug and through the EOS visit will be considered a concomitant medication

SECONDARY OUTCOMES:
Pharmacokinetics for primary cannabinoids and metabolites in Cohorts A and B: Cmin | Up to 21 days
  Minimum observed plasma concentration (Cmin)
Pharmacokinetics for primary cannabinoids and metabolites in Cohorts A and B: Cmax | Up to 21 days
  Maximum observed plasma concentration (Cmax)
Pharmacokinetics for primary cannabinoids and metabolites in Cohorts A and B: Tmax | Up to 21 days
  Time of maximum serum concentration (Tmax)
Pharmacokinetics for primary cannabinoids and metabolites in Cohort A: AUC0-last | Up to 21 days
  Area under the plasma concentration-time curve from time zero to the last quantifiable time point (AUC0-last)
Pharmacokinetics for primary cannabinoids and metabolites in Cohort A: AUC0-inf | Up to 21 days
  Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-inf) [including percent of area under the curve obtained by extrapolation (AUCExtrap)]
Pharmacokinetics for primary cannabinoids and metabolites in Cohorts A and B: lz | Up to 21 days
  Terminal rate constant (lz)
Pharmacokinetics for primary cannabinoids and metabolites in Cohorts A and B: t1/2 | Up to 21 days
  Half-life (t1/2)
Pharmacokinetics for primary cannabinoids and metabolites in Cohort A: Cl/F | Up to 21 days
  Apparent clearance (Cl/F)
Pharmacokinetics for primary cannabinoids and metabolites in Cohort A: Vz/F | Up to 21 days
  Apparent volume of distribution (Vz/F)
Pharmacokinetics for primary cannabinoids and metabolites in Cohort A: CTlast | Up to 21 days
  Concentration at last time point (CTlast)
Pharmacokinetics for primary cannabinoids and metabolites in Cohort B: AUC0-tau | Up to 21 days
  Area under the concentration-time curve from time zero to the end of the dosing interval (tau) at steady state (AUC0-tau)
Pharmacokinetics for primary cannabinoids and metabolites in Cohort B: Vd/F,ss | Up to 21 days
  Apparent volume of distribution at steady state (Vd/F,ss)
Pharmacokinetics for primary cannabinoids and metabolites in Cohort B: Cl/F,ss | Up to 21 days
  Apparent clearance at steady state (Cl/F,ss)
Pharmacokinetics for primary cannabinoids and metabolites in Cohort B: Aer | Up to 21 days
  Cumulative amount excrete renally (Aer)
Pharmacokinetics for primary cannabinoids and metabolites in Cohort B: fe% | Up to 21 days
  Fraction of unchanged drug excreted (fe%)
Pharmacokinetics for primary cannabinoids and metabolites in Cohort B: CLr [Ae0-t/AUC0-t] | Up to 21 days
  Renal clearance (CLr [Ae0-t/AUC0-t])
Change from baseline in subjective pharmacodynamic effects | Up to 21 days
  Assessed using the Drug Effects Questionnaire, a validated instrument commonly used in psychoactive drug research consisting of 20 items that are each rated using a unipolar 100 mm visual analog scale, with anchors of "not at all" on one end and "extremely" on the other. Participants are instructed to rate how they were feeling "right now" on six items related to the investigational study product: feeling the effect, liking any of the effects, disliking any of the effects, feeling any good effects, feeling any bad effects and likelihood of taking the study product again. Additionally, participants rate how much they are experiencing the following 14 adjectives: "sick," "heart racing," "anxious," "relaxed," "paranoid," "tired/drowsy," "alert," "irritable," "energetic," "restless," "hungry," "dazed," "distracted" and "euphoric/happy."

CONTACTS AND LOCATIONS:
Overall Officials: Kristi McLendon, MD, Principal Investigator — Q-Pharm Pty Ltd
Locations (1):
- Q-Pharm Pty Ltd, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No